CLINICAL TRIAL: NCT03880474
Title: A Phase 2b Study to Determine the Efficacy of Candidate Influenza Vaccine MVA-NP+M1 in Adults Aged 18 Years and Over
Brief Title: Efficacy of Candidate Influenza Vaccine MVA-NP+M1 in Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial is being stopped for futility. Season 2 cancelled.
Sponsor: Barinthus Biotherapeutics (Industry)
Collaborators: Clinical Network Services (CNS) Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FLU009
Record Dates: First submitted 2019-02-21; First posted 2019-03-19 (Actual); Results first posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MVA-NP+M1 (Experimental): Vaccination administered: MVA-NP+M1 (IM injection, 0.5 ml, 1.5 x10^8 pfu.)
  Interventions: Biological: MVA-NP+M1
- Saline Placebo (Placebo Comparator): Vaccination administered: Sodium Chloride (IM injection, 0.5 ml, 0.9%)
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: MVA-NP+M1 — Trial Vaccine
  Arms: MVA-NP+M1
Drug: Saline — Sodium Chloride Placebo
  Other Names: Placebo
  Arms: Saline Placebo

SUMMARY:
A Phase 2b Study to Determine the Efficacy of Candidate Influenza Vaccine MVA-NP+M1 in Adults aged 18 years and over. To assess the effect of MVA-NP+M1 on the reduction of laboratory confirmed influenza when given as an adjunct to licensed quadrivalent influenza vaccine (QIV) in adults

DETAILED DESCRIPTION:
This is a Phase 2b, multicentre, randomised, single-blind study in up to 6000 adults to compare the efficacy, safety and immunogenicity of MVA-NP+M1 when given as an adjunct to a standard, licensed adult dose of QIV. The study will be conducted on an outpatient basis and will run over two consecutive influenza seasons. It is aimed to recruit 2200 participants in Season 1 and 2800-3800 participants in Season 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults aged 18 years and over
* Receipt of a standard-dose licensed influenza QIV vaccine on the day of, or within 28 days prior to, randomisation
* A female participant is eligible for this study if she is not pregnant or breast feeding and one of the following:

  1. Of non-childbearing potential (i.e. women who have had a hysterectomy or tubal ligation or are postmenopausal, as defined by no menses in greater than or equal to 1 year)
  2. Of childbearing potential but agrees to practice effective contraception 8 weeks post-vaccination and has a negative urine pregnancy test pre-vaccination. Acceptable methods of contraception include one or more of the following:

  i. Male partner who is sterile prior to the female participant's entry into the study and is the sole sexual partner for the female participant ii. Implants of levonorgestrel iii. Injectable progestogen iv. An intrauterine device with a documented failure rate of <1% v. Oral contraceptives vi. Double barrier methods including diaphragm or condom vii. Abstinence as long as it is line with the usual and preferred lifestyle of the participant
* Participant is willing and has capacity to provide written informed consent for participation in the study (in the Investigator's opinion)
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the Investigators to discuss the participant's medical history with their healthcare provider
* Present and able to visit the clinic in the event of an ILI episode during the influenza season

Exclusion Criteria:

* Any other significant disease, disorder or finding (including blood test results), which, in the opinion of the Investigator, would either put the participant at risk because of participation in the study, or may influence the result of the study
* Receipt of any investigational product within 6 months prior to study, or prior participation in a clinical study of any Influenza vaccine and agreement not to participate in another clinical study for the duration of study follow-up
* Prior receipt of an investigational vaccine likely to impact on interpretation of the study data
* Active infection with HIV, Hepatitis B or Hepatitis C (from patient history or medical records)
* History of severe allergic reactions (e.g. anaphylaxis)
* History of auto-immune disease e.g. Guillain-Barré syndrome
* Not willing to comply with study procedures
* Immunosuppressed or taking immunosuppressive medications
* Use of warfarin or other blood thinning medications (aspirin is acceptable)
* Tattoos or birthmarks at the vaccination site
* Participant bruises easily, has haematoma or keloid scarring
* Receipt of a licenced inactivated vaccine (e.g. pneumococcal vaccine) within 2 weeks prior to vaccination
* Receipt of an off licensed live vaccine (e.g. herpes zoster vaccine) within 4 weeks prior to vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2364 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Vandeleur, MD, Principal Investigator — Paratus Clinical Pty Ltd
Locations (9):
- Australia (9):
  - Paratus Clinical Pty Ltd, Blacktown, New South Wales
  - Genesis Research Services, Broadmeadow, New South Wales
  - Paratus Clinical Pty Ltd, Kanwal, New South Wales
  - Scientia Clinical Research, Sydney, New South Wales
  - University of Sunshine Coast (USC), Morayfield, Queensland
  - University of Sunshine Coast (USC), Sippy Downs, Queensland
  - Mater Research, South Brisbane, Queensland
  - CMAX, Adelaide, South Australia
  - Nucleus Network Pty Ltd, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evans TG, Bussey L, Eagling-Vose E, Rutkowski K, Ellis C, Argent C, Griffin P, Kim J, Thackwray S, Shakib S, Doughty J, Gillies J, Wu J, Druce J, Pryor M, Gilbert S. Efficacy and safety of a universal influenza A vaccine (MVA-NP+M1) in adults when given after seasonal quadrivalent influenza vaccine immunisation (FLU009): a phase 2b, randomised, double-blind trial. Lancet Infect Dis. 2022 Jun;22(6):857-866. doi: 10.1016/S1473-3099(21)00702-7. Epub 2022 Mar 16. PMID 35305317

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The single-blind study was conducted at 9 sites across Australia, over one Influenza season.
Pre-assignment Details: 2364 were screened and 2152 participants started randomized in a 1:1 ratio and received (along with a licensed adult dose of QIV), either active drug (MVA-NP+M1) or Placebo, via IM injection. Overall, 1077 participants received active drug and 1075 Placebo. A total of 2109 participants completed the study. The Immunogenicity Cohort was a subset of 50 participants: 25 participants were administered active drug and 25 participants were administered Placebo. All 50 participants completed the study.
Groups:
- MVA-NP+M1 Group (Main Cohort + Immunogenicity Cohort): Vaccination administered: 1 dose of MVA-NP+M1 (IM injection, 0.5 ml, 1.5 x10^8 pfu per dose) MVA-NP+M1: Trial Vaccine Vaccinations were administered by intramuscular injection on Day 0. The participants were provided with an oral thermometer, tape measure and electronic diary card (eDiary) and instructed how to complete the eDiary at home.
  Participants recorded their oral temperature and any solicited adverse events for 7 days post-vaccination and unsolicited adverse events for 28 days post-vaccination.
  The study team contacted participants by telephone on Day 1 (+2 days) post-vaccination and Day 7 (+3 days) post-vaccination for safety follow-up. If the participant had persistent, vaccine-related Grade 3 AEs during the first 4 weeks post-vaccination they could be asked to attend a further clinical assessment.
  The Immunogenicity Cohort of the MVA-NP+M1 group (25 participants), had pre vaccination safety laboratory and immunogenicity blood samples taken.
  In addition to the visits and procedures outlined above these participants attended an additional three clinic visits on Days 7 (+3 days), 28 (±7 days) and Week 26 (±1 week) (approximate end of the influenza season).
  At the end of the influenza season, all participants were contacted by telephone to inform them of the end of the follow-up period and confirm all information had been collected.
- Saline Placebo Group (Main Cohort+ Immunogenicity Cohort): Vaccination administered: 1 dose of Sodium Chloride (IM injection, 0.5 ml, 0.9% per dose) Saline: Sodium Chloride Placebo Vaccinations were administered by intramuscular injection on Day 0. The participants were provided with an oral thermometer, tape measure and electronic diary card (eDiary) and instructed how to complete the eDiary at home.
  Participants recorded their oral temperature and any solicited adverse events for 7 days post-vaccination and unsolicited adverse events for 28 days post-vaccination.
  The study team contacted participants by telephone on Day 1 (+2 days) post-vaccination and Day 7 (+3 days) post-vaccination for safety follow-up. If the participant had persistent, vaccine-related Grade 3 AEs during the first 4 weeks post-vaccination they could be asked to attend a further clinical assessment.
  The Immunogenicity Cohort of the Placebo group (25 participants), had pre vaccination safety laboratory and immunogenicity blood samples taken.
  In addition to the visits and procedures outlined above these participants attended an additional three clinic visits on Days 7 (+3 days), 28 (±7 days) and Week 26 (±1 week) (approximate end of the influenza season).
  At the end of the influenza season, all participants were contacted by telephone to inform them of the end of the follow-up period and confirm all information had been collected.
Period: Overall Study
Arm/Group | MVA-NP+M1 Group (Main Cohort + Immunogenicity Cohort) | Saline Placebo Group (Main Cohort+ Immunogenicity Cohort)
Started | 1077 | 1075
Completed | 1054 | 1055
Not Completed | 23 | 20

BASELINE CHARACTERISTICS:
Groups:
- MVA-NP+M1 Group: Vaccination administered: 1 dose of MVA-NP+M1 (IM injection, 0.5 ml, 1.5 x10^8 pfu per dose) MVA-NP+M1: Trial Vaccine Vaccinations were administered by intramuscular injection on Day 0. The participants were provided with an oral thermometer, tape measure and electronic diary card (eDiary) and instructed how to complete the eDiary at home.
  Participants recorded their oral temperature and any solicited adverse events for 7 days post-vaccination and unsolicited adverse events for 28 days post-vaccination.
  The study team contacted participants by telephone on Day 1 (+2 days) post-vaccination and Day 7 (+3 days) post-vaccination for safety follow-up. If the participant had persistent, vaccine-related Grade 3 AEs during the first 4 weeks post-vaccination they could be asked to attend a further clinical assessment.
  The Immunogenicity Cohort of the MVA-NP+M1 group (25 participants), had pre vaccination safety laboratory and immunogenicity blood samples taken.
  In addition to the visits and procedures outlined above these participants attended an additional three clinic visits on Days 7 (+3 days), 28 (±7 days) and Week 26 (±1 week) (approximate end of the influenza season).
  At the end of the influenza season, all participants were contacted by telephone to inform them of the end of the follow-up period and confirm all information had been collected.
- Saline Placebo Group: Vaccination administered: 1 dose of Sodium Chloride (IM injection, 0.5 ml, 0.9% per dose) Saline: Sodium Chloride Placebo Vaccinations were administered by intramuscular injection on Day 0. The participants were provided with an oral thermometer, tape measure and electronic diary card (eDiary) and instructed how to complete the eDiary at home.
  Participants recorded their oral temperature and any solicited adverse events for 7 days post-vaccination and unsolicited adverse events for 28 days post-vaccination.
  The study team contacted participants by telephone on Day 1 (+2 days) post-vaccination and Day 7 (+3 days) post-vaccination for safety follow-up. If the participant had persistent, vaccine-related Grade 3 AEs during the first 4 weeks post-vaccination they could be asked to attend a further clinical assessment.
  The Immunogenicity Cohort of the Placebo group (25 participants), had pre vaccination safety laboratory and immunogenicity blood samples taken.
  In addition to the visits and procedures outlined above these participants attended an additional three clinic visits on Days 7 (+3 days), 28 (±7 days) and Week 26 (±1 week) (approximate end of the influenza season).
  At the end of the influenza season, all participants were contacted by telephone to inform them of the end of the follow-up period and confirm all information had been collected.
- Total: Total of all reporting groups
Arm/Group | MVA-NP+M1 Group | Saline Placebo Group | Total
Number analyzed (Participants) | 1077 | 1075 | 2152
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (18.93) | 43.8 (18.40) | 43.7 (18.66)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 631 | 631 | 1262
  Male | 445 | 443 | 888
  Unknown | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 21
  Not Hispanic or Latino | 1061 | 1052 | 2113
  Unknown or Not Reported | 6 | 12 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 143 | 118 | 261
  Native Hawaiian or Other Pacific Islander | 8 | 13 | 21
  Black or African American | 9 | 7 | 16
  White | 882 | 892 | 1774
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 29 | 42 | 71
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.36 (6.727) | 28.26 (6.143) | 28.31 (6.435)
Body Temperature [Mean (Standard Deviation); unit: degree Celsius] | 36.44 (0.420) | 36.44 (0.401) | 36.44 (0.410)

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Laboratory Confirmed Influenza Using Reverse Transcription Polymerase Chain Reaction (RT-PCR).
Description: The measure used reverse transcription polymerase chain reaction (RT-PCR) on deep nasal/mid-turbinate swab samples to record confirmed cases of influenza.
  If influenza symptoms are experienced at any time during the Follow Up period, after the vaccination, participants will attend the clinic on two occasions, the first as soon as possible and at least within 72 hours of the onset of symptoms for deep nasal swabs to be taken. Both swabs must be taken within 96 hours of symptom onset.
  The incidence rate of laboratory confirmed influenza using RT-PCR will be estimated for each vaccine group. The 95% CI for the incidence rate will be estimated by mid-p exact method. The difference in incidence rate between vaccine groups will be compared by Fisher's exact method.
Time Frame: 210 days (during the influenza season, starting on 01 May 2019 and ending on or before 15 October 2019) in line with official Australian influenza season.
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-NP+M1 Group | Saline Placebo Group
Number analyzed (Participants) | 1077 | 1075
Participants
  Participants with laboratory confirmed influenza using RT-PCR | 35 | 23
  Participants without laboratory confirmed influenza using RT-PCR | 1042 | 1052
Statistical Analysis 1: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Test type: Other; p = 0.1146, Log Binominal Model; Relative Risk = 1.52, 95% CI 2-sided [0.90 to 2.55]
Statistical Analysis 2: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Test type: Other; p = 0.1146, Poisson Model with Robust Variance; Relative Risk = 1.52, 95% CI 2-sided [0.90 to 2.55]

2. Secondary Outcome: Number and Percentage of Participants With Influenza-like Illness (ILI) as Derived From Daily ILI eDiary
Description: ILI is defined as feeling feverish or having a fever (feeling feverish or having a fever (≥37.8Celsius)) and at least one of the following symptoms: cough, sore throat.
  The incidence rate of ILI by the participant completing of eDiaries will be estimated for each vaccine group. The 95% CI for the incidence will be estimated by mid-p exact method. The difference in incidence between groups will be compared by Fisher's exact method.
Time Frame: 210 days (during the influenza season, starting on 01 May 2019 and ending on or before 15 October 2019)
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-NP+M1 Group | Saline Placebo Group
Number analyzed (Participants) | 1077 | 1075
Participants
  Positive ILI Cases | 273 | 273
  Negative ILI Cases | 804 | 802
Statistical Analysis 1: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; The Analysis concerns the Incidence of Influenza-like Illness (ILI); Test type: Other; p = 1.0000, Log Binomial Model; Relative Risk = 1, 95% CI 2-sided [0.86 to 1.15]
Statistical Analysis 2: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; The Analysis concerns the Incidence of Influenza-like Illness (ILI); Test type: Other; p = 0.9799, Poisson Model with Robust Variance; Relative Risk = 1, 95% CI 2-sided [0.86 to 1.15]

3. Secondary Outcome: Number and Percentage of Participants With Solicited Local and Systemic Reactogenicity Signs and Symptoms for 7 Days Following Vaccination (and Occurrence of Serious Adverse Events SAEs)
Description: The solicited adverse events are commonly observed soon after receipt of vaccines and relate to local and systemic signs and symptoms.
  The solicited local injection site reactions (ISR) include pain, induration, warmth, and erythema (redness).
  The solicited systemic reactions include feverishness, chills, myalgia, fatigue, headache, nausea, arthralgia, and malaise.
  Participants completed eDiaries post vaccination to record ISR and systemic reactogenicity over the first 7 days post-vaccination (and the ongoing (S)AEs throughout the study).
  The participant reporting of all ISR categories and solicited systemic reactions was compared between the MVA-NP+M1 treated group and the Placebo treated group.
  Diary reported ISRs and solicited systemic reactions were summarized, by vaccination group, using descriptive statistics.
Time Frame: 7 days to a total of 210 days for SAEs (over the duration of the influenza season, between 01 May and 15 October)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-NP+M1 Group | Saline Placebo Group
Number analyzed (Participants) | 1077 | 1075
Participants
  Participants with Solicited Local Injection Site Reaction (IRS) - Pain | 292 | 19
  Participants with Solicited Local Injection Site Reaction (IRS) - Induration | 113 | 4
  Participants with Solicited Local Injection Site Reaction (IRS) - Warmth | 205 | 18
  Participants with Solicited Local Injection Site Reaction (IRS) - Erythema | 198 | 15
  Participants with Severe, Solicited Local Injection Site Reaction | 12 | 1
  Participants with Solicited Systemic Reactions - Chills | 61 | 18
  Participants with Solicited Systemic Reactions - Myalgia | 256 | 85
  Participants with Solicited Systemic Reactions - Fatigue | 248 | 117
  Participants with Solicited Systemic Reactions - Headache | 238 | 106
  Participants with Solicited Systemic Reactions - Nausea | 88 | 31
  Participants with Solicited Systemic Reactions - Arthralgia | 156 | 57
  Participants with Solicited Systemic Reactions - Malaise | 273 | 139
  Participants with Solicited Systemic Reactions - Feverishness | 214 | 93
  Participants with Severe, Solicited Systemic Reaction | 45 | 14

4. Secondary Outcome: Number of Participants With Immunogenic Response (Immunogenicity of MVA-NP+M1 in Adjunction With Licensed QIV as Assessed Via Titres of Influenza-specific Neutralizing Antibodies)
Description: The numbers of Immunogenic Participants (participants with positive immune response as assessed at Day 28 and week 26 in relation to the baseline day 0 Immunogenicity) were summarized and listed.
  The immunogenicity here was assessed as the geometric mean titers of influenza-specific neutralizing antibodies at different timepoints in relation to the baseline, against the antigens included in the licensed QIV(Influenza A/H3N2 (HI), Influenza A/H3N2 (MN), Influenza A/H3N2 (H1N1pdm), Influenza B/Victoria, and Influenza B/Yamagata).
  The neutralizing antibody assays included microneutralisation and hemagglutination inhibition titers using standard methodologies for the four strains that were in the licensed vaccine.
  The immunogenicity analyses were conducted only on the Immunology Analysis Set of Participants.
Time Frame: Day 28 and Week 26
Population: The samples for immunogenicity analysis were taken only from participants in the 2 Immunogenicity cohorts included in the MVA-NP+M1 Group vs the Placebo Group.
  The immunogenicity analysis for Day 28 used a number of 24 participant results from the MVA-NP+M1 Cohort and a number of 24 participant results from the Placebo Cohort.
  The immunogenicity analysis for Week26 used a number of 23 participant results from the MVA-NP+M1 Cohort and a number of 25 participant results from the Placebo Cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-NP+M1 Group | Saline Placebo Group
Number analyzed (Participants) | 25 | 25
Participants
  Participants with Influenza Antibody Titer: ANCOVA Analysis Immunology, at Day 28: number analyzed (Participants) | 24 | 24
  Participants with Influenza Antibody Titer: ANCOVA Analysis Immunology, at Day 28 | 23 | 24
  Participants with Influenza Antibody Titer: ANCOVA Analysis Immunology, at Week 26: number analyzed (Participants) | 23 | 25
  Participants with Influenza Antibody Titer: ANCOVA Analysis Immunology, at Week 26 | 23 | 25
Statistical Analysis 1: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Titers of influenza-specific neutralizing antibodies against Influenza A/H3N2 (HI) at Day 28; Test type: Other; p = 0.3284, ANCOVA; Least Squares Mean Difference = -287.1, 95% CI 2-sided [-872.75 to 298.59]
Statistical Analysis 2: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Titers of influenza-specific neutralizing antibodies against Influenza A/H3N2 (HI) at Week26; Test type: Other; p = 0.8468, ANCOVA; Least Squares Mean Difference = -13.39, 95% CI 2-sided [-152.26 to 125.47]
Statistical Analysis 3: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Titers of influenza-specific neutralizing antibodies against Influenza A/H3N2 (MN) at Day 28; Test type: Other; p = 0.5087, ANCOVA; Least Squares Mean Difference = -465.7, 95% CI 2-sided [-1875.21 to 943.75]
Statistical Analysis 4: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Titers of influenza-specific neutralizing antibodies against Influenza A/H3N2 (MN) at Week 26; Test type: Other; p = 0.7509, ANCOVA; Least Squares Mean Difference = -83.68, 95% CI 2-sided [-611.67 to 444.32]
Statistical Analysis 5: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Titers of influenza-specific neutralizing antibodies against Influenza A/H1N1pdm at Day 28; Test type: Other; p = 0.3398, ANOVA; Least Squares Mean Difference = -81.17, 95% CI 2-sided [-250.72 to 88.39]
Statistical Analysis 6: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Titers of influenza-specific neutralizing antibodies against Influenza A/H1N1pdm at Week 26; Test type: Other; p = 0.4154, ANCOVA; Least Squares Mean Difference = 26.15, 95% CI 2-sided [-37.95 to 90.26]
Statistical Analysis 7: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Titers of neutralizing antibodies against Influenza B/ Victoria at Day 28; Test type: Other; p = 0.7193, ANCOVA; Least Squares Mean Difference = 22.84, 95% CI 2-sided [-104.50 to 150.18]
Statistical Analysis 8: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Titers of influenza-specific neutralizing antibodies against Influenza B/ Victoria at Week 26; Test type: Other; p = 0.1496, ANCOVA; Least Squares Mean Difference = 52.38, 95% CI 2-sided [-19.59 to 124.35]
Statistical Analysis 9: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Titers of influenza-specific neutralizing antibodies against Influenza B/Yamagata at Day 28; Test type: Other; p = 0.9044, ANCOVA; Least Squares Mean Difference = -16.76, 95% CI 2-sided [-296.57 to 263.06]
Statistical Analysis 10: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Titers of influenza-specific neutralizing antibodies against Influenza B/Yamagata at Week 26; Test type: Other; p = 0.4198, ANCOVA; Least Squares Mean Difference = 38.64, 95% CI 2-sided [-56.97 to 134.24]

5. Secondary Outcome: Duration of Influenza-like Illness (ILI) as Derived From Daily ILI eDiary
Description: The duration of ILI is defined as the duration (days) from the first day ILI criteria met (as defined at the Secondary Outcome Measure 2) until the first day afterwards ILI criteria not met (event, ILI recovery).
  ILI positive participants with ILI criteria met throughout the entire influenza season were censored at the last day recorded with the ILI dairy.
  Survival analysis was used for the analysis of duration of ILI. The survival function for the duration of ILI was estimated by the Kaplan-Meier method.
Time Frame: 210 days (during the influenza season, starting on 01 May 2019 and ending on or before 15 October 2019)
Population: ILI duration analysis is only applicable for ILI positive participants. In the MVA-NP+M1 Group there were 273 ILI positive participants assessed: 247 with event and 26 censored; In the Placebo Group there were 273 ILI positive participants assessed: 248 with event and 25 censored.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | MVA-NP+M1 Group | Saline Placebo Group
Number analyzed (Participants) | 273 | 273
days | 3 [3 to 4] | 3 [3 to 4]
Statistical Analysis 1: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Test type: Other; p = 0.4159, Regression, Cox; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.90 to 1.28]

6. Secondary Outcome: Severity of Influenza-like Illness (ILI) Derived From Daily ILI eDiary as Time Weighted AUC
Description: The severity of ILI was assessed by each participant completing of electronic Diaries for symptom severity daily for the following symptoms: Feeling hot, Temperature, Cough, Sore throat, Blocked nose, Chest pain, Muscle aches, Shortness of breath with their severities (scores) recorded as: Not Present (0), Mild (1), Moderate (2), Severe (3). For each symptom, the severity score was used to calculate the area under the curve (AUC), along with the calendar day, for the entire influenza season using trapezoidal rule. Participants could be followed for varying days in the influenza season, therefore the AUC will be time weighted to 168 days: Time weighted AUC=((raw AUC [time in days])/(number of days used for analysis)) * 168
Time Frame: 210 days (during the influenza season, starting on 01 May 2019 and ending on or before 15 October 2019)
Measure: Mean (Standard Deviation); unit: weighted days
Arm/Group | MVA-NP+M1 Group | Saline Placebo Group
Number analyzed (Participants) | 1077 | 1075
weighted days | 5490 (23.4944) | 5297 (21.3996)
Statistical Analysis 1: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Time Weight Area Under the Curve (AUC) for Symptoms of Influenza - Symptom: Feeling Hot (AUC); Test type: Other; p = 0.9550, ANOVA; Geometric Mean Ratio (Active vs Placebo) = 0.99, 95% CI 2-sided [0.83 to 1.19]
Statistical Analysis 2: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Time Weight Area Under the Curve (AUC) for Symptoms of Influenza - Symptom: Temperature (AUC); Test type: Other; p = 0.8933, ANOVA; Geometric Mean Ratio (Active vs Placebo) = 1, 95% CI 2-sided [1 to 1]
Statistical Analysis 3: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Time Weight Area Under the Curve (AUC) for Symptoms of Influenza - Symptom: Cough (AUC); Test type: Other; p = 0.2156, ANOVA; Geometric Mean Ratio (Active vs Placebo) = 0.87, 95% CI 2-sided [0.7 to 1.09]
Statistical Analysis 4: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Time Weight Area Under the Curve (AUC) for Symptoms of Influenza - Symptom: Sore Throat AUC; Test type: Other; p = 0.2216, ANOVA; Geometric Mean Ratio (Active vs Placebo) = 0.88, 95% CI 2-sided [0.71 to 1.10]
Statistical Analysis 5: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Time Weight Area Under the Curve (AUC) for Symptoms of Influenza - Symptom: Blocked Nose AUC; Test type: Other; p = 0.2306, ANOVA; Geometric Mean Ratio (Active vs Placebo) = 0.87, 95% CI 2-sided [0.69 to 1.09]
Statistical Analysis 6: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Time Weight Area Under the Curve (AUC) for Symptoms of Influenza - Symptom: Chest Pain AUC; Test type: Other; p = 0.8038, ANOVA; Geometric Mean Ratio (Active vs Placebo) = 0.99, 95% CI 2-sided [0.97 to 1.13]
Statistical Analysis 7: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Time Weight Area Under the Curve (AUC) for Symptoms of Influenza - Symptom: Muscle Pain AUC; Test type: Other; p = 0.9319, ANOVA; Geometric Mean Ratio (Active vs Placebo) = 1.01, 95% CI 2-sided [0.84 to 1.21]
Statistical Analysis 8: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Time Weight Area Under the Curve (AUC) for Symptoms of Influenza - Symptom: Shortness of Breath AUC; Test type: Other; p = 0.8399, ANOVA; Geometric Mean Ratio (Active vs Placebo) = 1.01, 95% CI 2-sided [0.86 to 1.19]

7. Secondary Outcome: Number of Participants With Immunogenic Response to MVA-NP+M1 (as Assessed Via the Frequency of Influenza-specific T-cells)
Description: The numbers of immunogenic Participants (with positive immune response as assessed at Day 28 and week 26 in relation to the baseline day 0 Immunogenicity) were listed.
  The immunogenicity here was determined via the frequency of influenza-specific T-cells measured by IFN-γ/granzyme B ELISpot assay (enzyme linked immunospot) where the adjusted Spot Forming Units (SFU) per million PBMCs (peripheral blood mononuclear cells) after background subtraction (dimethyl sulfoxide, DMSO) were counted.
  The immunogenicity analyses were conducted only in the Immunology Analysis Set of Participants.
Time Frame: Day 28 and Week 26
Population: The samples for this immunogenicity analysis were taken only from participants in the 2 Immunogenicity cohorts included in the MVA-NP+M1 Group vs the Placebo Group.
  The immunogenicity analysis for Day 28 used 24 participant results from the MVA-NP+M1 Cohort and 24 participant results from the Placebo Cohort, as available.
  The immunogenicity analysis for Week26 used 23 participant results from the MVA-NP+M1 Cohort and 25 participant results from the Placebo Cohort, as available.
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-NP+M1 Group | Saline Placebo Group
Number analyzed (Participants) | 25 | 25
Participants
  Participants with immunogenic response (as the frequency of influenza-specific T-cells) at Day 28: number analyzed (Participants) | 24 | 24
  Participants with immunogenic response (as the frequency of influenza-specific T-cells) at Day 28 | 20 | 21
  Participants with Immunogenic response (via the frequency of influenza-specific T-cells) at Week 26: number analyzed (Participants) | 23 | 25
  Participants with Immunogenic response (via the frequency of influenza-specific T-cells) at Week 26 | 16 | 13
Statistical Analysis 1: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Statistical analysis was performed for Total(NP+M) (SFU/10^6 PBMC) at Day 28 Nucleoprotein = NP, matrix1 = M1; Test type: Other; p = 0, ANCOVA; Least Squares Mean Difference = 743.78, 95% CI 2-sided [443.71 to 1043.84]
Statistical Analysis 2: Comparison: MVA-NP+M1 Group vs Saline Placebo Group; Statistical analysis was performed for Total(NP+M) (SFU/10^6 PBMC) at Week 26 Nucleoprotein = NP, matrix1 = M1; Test type: Other; p = 0.0673, ANCOVA; Least Squares Mean Difference = 177.10, 95% CI 2-sided [-13.14 to 367.33]

ADVERSE EVENTS:
Time Frame: Unsolicited non-serious adverse events will be collected for 28 days post-vaccination. Hospitalisations, other serious adverse events and or adverse events of special interest will be collected for the duration of the influenza season. Solicited adverse events, including solicited local injection site reactions (ISR) and solicited systemic reactions, will be collected for 7 days post-vaccination. These will be recorded daily in the eDiary for all participants.
Description: Adverse events were coded using MedDRA(most recent version). AEs are grouped by system organ class (SOC) and preferred term and summarized by vaccination group (MVA-NP+M1 Group vs Saline Placebo Group) at the time of AE onset. All AEs are reported for each group and the Immunogenicity cohorts (as parts of each group) did not influence the adverse events reporting style.
  In the summary tables, adverse events are presented/summarized by decreasing frequency of Total Events overall within each SOC
Arm/Group | MVA-NP+M1 Group | Saline Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/1077 | 1/1075
Serious Adverse Events (participants affected / at risk) | 18/1077 | 22/1075
Other Adverse Events (participants affected / at risk) | 524/1077 | 435/1075
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVA-NP+M1 Group (N=1077) | Saline Placebo Group (N=1075)
Pneumonia (Infections and infestations) | 2 (3) | 3 (3)
Diverticulitis (Infections and infestations) | 1 (1) | 1
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Medical device site joint infection (Immune system disorders) | 1 (1) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Endometriosis ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Adnexal torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVA-NP+M1 Group (N=1077) | Saline Placebo Group (N=1075)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 115 (122) | 119 (127)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 89 (97) | 93 (102)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 90 (95) | 84 (93)
Cough (Respiratory, thoracic and mediastinal disorders) | 73 (76) | 86 (91)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 25 (28) | 12 (13)
Headache (Nervous system disorders) | 145 (170) | 122 (135)
Dizziness (Nervous system disorders) | 12 (12) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 12 (15)
Injection site pain (General disorders) | 73 (74) | 0 (0)
Fatigue (General disorders) | 43 (46) | 24 (25)
Pyrexia (General disorders) | 30 (32) | 0 (0)
Malaise (General disorders) | 16 (18) | 19 (21)
Influenza like illness (General disorders) | 23 (23) | 15 (15)
Feeling hot (General disorders) | 11 (11) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 59 (61) | 36 (39)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (12) | 13 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 11 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (11) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 20 (22) | 31 (34)
Nasopharyngitis (Infections and infestations) | 12 (12) | 15 (16)
Influenza (Infections and infestations) | 11 (11) | 0 (0)
Nausea (Gastrointestinal disorders) | 26 (28) | 24 (26)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 15 (16)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS (Injury, poisoning and procedural complications) | 25 (30) | 24 (27)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 19 (22) | 18 (19)
Seasonal allergy (Immune system disorders) | 14 (15) | 12 (14)
EAR AND LABYRINTH DISORDERS (Ear and labyrinth disorders) | 14 (15) | 12 (12)
EYE DISORDERS (Eye disorders) | 0 (0) | 14 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT03880474/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT03880474/SAP_001.pdf